CLINICAL TRIAL: NCT04893668
Title: Depression and Anxiety in Long Term COVID 19. A Study in Neurotransmitter Impact of Severe Acute Respiratory Syndrome-Coronavirus 2 Infection.
Brief Title: Depression and Anxiety in Long Term Coronavirus Disease COVID-19
Acronym: DALT-COV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Other Study IDs: 1105211301
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Covid19; Depression; Anxiety
Keywords: Covid19; Serotonin; Dopamine; Depression; Anxiety
MeSH Terms: conditions — COVID-19; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood Sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed with COVID 19: The participant with confirmed RT-PCR Covid 19 at the beginning of the study
  Interventions: Other: Depression; Other: Anxiety
- Unexposed with COVID 19: The participant without confirmed RT-PCR Covid 19 at the beginning of the study until 6 month follow up period
  Interventions: Other: Depression; Other: Anxiety

INTERVENTIONS:
Other: Depression — Any participants who develop depression symptoms according to DSM 5 criteria
Other: Anxiety — Any participants who develop anxiety symptoms according to DSM 5 criteria

SUMMARY:
Background :

Depression and Anxiety are linked to COVID (Coronavirus Disease)-19 long-term impact through several mechanisms. The possible way is the alteration of neurotransmitter regulation from the interaction of severe acute respiratory syndrome -Coronavirus-2 (SARS-COV2) with Angiotensin-Converting Enzyme 2 (ACE2) receptor, and Dopa Decarboxylase (DDC), an enzyme that associated with the production of dopamine, serotonin, and other neurotransmitters. However, some arguments exist that depression and anxiety occur naturally due to external stressors, as the impact of public health measures, and not associated with physiological changes due to viral infection.

Objective:

1. This study aims to identify whether the patient discharged after COVID 19 treatment has significant changes in serotonin and dopamine level which might induce depression and anxiety internally and,
2. To distinguish external etiologies that might induce depression and anxiety such as social isolation and stress due to public health restriction.

Method:

A prospective longitudinal study of people with the interest exposure is COVID 19 and the primary outcome is Depression, Anxiety, and Neurotransmitter level

Hypothesis:

People with a previous infection of COVID 19 have a significant difference in neurotransmitter level over time and compared to non exposed group and a higher prevalence of anxiety and depression.

DETAILED DESCRIPTION:
Method :

Prospective Longitudinal study for 6 months. with both exposed and unexposed group

Target population :

A cohort of the population in multiple centers (3 centers)

Sample Size Calculation with Longitudinal study formula:

1. Effect Size: 0.15
2. Type I error: 0.05
3. Power of Study: 80%
4. Number of Group: 2
5. Repeated measurement: 3 times
6. Correlation among Repeated Measures: 0.5
7. Nonsphericity Correction: 1
8. Initial Sample size: 75

Adjusted by clustering effect:

1. Intraclass Correlation Coefficient = 0.05
2. Number of people per cluster = 25
3. Design Effect= 1 + 0.05(25-1) = 2.2
4. Total sample size = 75 x 2.2 = 165 participants

Procedure:

1. Participants will be assessed for eligibility
2. Screening for Depression, Anxiety, and Stress using Depression Anxiety Stress Scale (DASS) Questionnaire. Health-Related Quality of Life (QoL) and Pittsburgh Sleep Quality Index (PSQI)
3. Sample Collection and assessment of QoL, DASS, PSQI on the first day
4. Sample Collection and assessment of QoL, DASS, PSQI on day 60
5. Sample Collection and assessment of QoL, DASS, PSQI on day 120

Variables

1. Case Definition: Realtime Polymerase Chain Reaction (RT-PCR) and Cycle Threshold Value (CT)
2. Degree of COVID 19 Symptom-based on World Health Organization Criteria (Asymptomatic, Mild, Moderate, Severe, Critical)
3. Sociodemographic Variables (Age, Gender, Education, Income, Marital Status)
4. Sleep Quality using Pittsburgh Sleep Quality Index (PSQI)
5. Treatment of COVID: Antiviral, Antibiotic, Interleukin-6 Antagonist, Steroid, Plasma Convalescent, Ventilator, Human Intravenous Immunoglobulin, anticoagulant
6. Chronic Disease including Diabetes Mellitus, Hypertension, Chronic Kidney Disease
7. Medication that affects neurotransmitter level taken prior to recruitment.
8. History of Smoking classified by Brinkmann Index.
9. Body Mass Index
10. Complete Blood Count
11. Vaccination history

Outcome

1. Dopamine Serum
2. Serotonin Serum
3. Prevalence of Anxiety, and Depression according to Diagnostic and Statistical Manual of Mental disorders (DSM) 5

Statistical analysis Basic Analysis: Intention to Treat analysis

1. Linear Mixed Model for Neurotransmitter
2. Generalized Estimating Equation for Prevalence of Anxiety and Depression
3. Sensitivity analysis will be conducted, concerning the lost-to-follow up
4. A subgroup analysis will be conducted, particularly the participants with specific comorbidities

ELIGIBILITY:
Inclusion Criteria:

1. Age minimum 18 years old
2. For exposed group should be confirmed with RT-PCR
3. Not being diagnosed by depression or anxiety prior to recruitment

Exclusion Criteria:

1. The unexposed participants will be excluded from the unexposed group if contracted with the virus within the 6-month observation.
2. Patient falls into critical condition and it is unlikely to attend at least one follow-up measurement
3. Patient refuses to continue observation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three clusters will be appointed as the study center. The level of the cluster is at the municipality level where participants will be recruited consecutively
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Level of Serotonin | Changes of Serotonin level from the baseline to 60 days and 120 days
  The level of serotonin (5-hydroxytryptamine) measured from the blood serum with the normal range between 50 to 200 ng/mL
Level of Dopamine | Changes of Dopamine level from the baseline to 60 days and 120 days
  The level of serotonin (4- (2-aminoethyl) benzene-1, 2-diol) measured from the blood serum with the normal range between 0 to 30 pg/mL

SECONDARY OUTCOMES:
Prevalence of Depression | changes of prevalence of depression from the baseline to 60 days and 120 days
  Prevalence of depression defined in Diagnostic and Statistical Manual of Mental disorders fifth edition / DSM 5
Prevalence of Anxiety | changes of prevalence of Anxiety from the baseline to 60 days and 120 days
  Prevalence of Anxiety defined in Diagnostic and Statistical Manual of Mental disorders fifth edition / DSM 5

CONTACTS AND LOCATIONS:
Overall Officials: Bumi Herman, M.D Ph.D, Principal Investigator — Chulalongkorn University
Locations (1):
- Hasanuddin University Medical Research Center / HUMRC, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Protocol, Statistical Analysis Plan and De-identified data will be shared accordingly

REFERENCES:
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] Nataf S. An alteration of the dopamine synthetic pathway is possibly involved in the pathophysiology of COVID-19. J Med Virol. 2020 Oct;92(10):1743-1744. doi: 10.1002/jmv.25826. Epub 2020 Apr 8. No abstract available. PMID 32246784
- [Background] Antonini A, Leta V, Teo J, Chaudhuri KR. Outcome of Parkinson's Disease Patients Affected by COVID-19. Mov Disord. 2020 Jun;35(6):905-908. doi: 10.1002/mds.28104. Epub 2020 May 28. No abstract available. PMID 32347572
- [Background] Adhanom Ghebreyesus T. Addressing mental health needs: an integral part of COVID-19 response. World Psychiatry. 2020 Jun;19(2):129-130. doi: 10.1002/wps.20768. No abstract available. PMID 32394569
- [Background] Basagana X, Xiaomei Liao, Spiegelman D. Power and sample size calculations for longitudinal studies estimating a main effect of a time-varying exposure. Stat Methods Med Res. 2011 Oct;20(5):471-87. doi: 10.1177/0962280210371563. Epub 2010 Jun 14. PMID 20547587